CLINICAL TRIAL: NCT06460259
Title: The Effect of Breathing Exercises on Pain, Anxiety, Dyspnea, and Insomnia in Patients Undergoing Lung Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Fatma Gündoğdu, Principal Investigator, Assistant Professor, PhD, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2023/026
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Lung Surgery
Keywords: Breathing exercises; Insomnia; Pain; Anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain; Anxiety Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patients undergoing VATS or wedge resection procedures will be informed and their consent will be obtained prior to the procedure. Individuals who consent and meet the inclusion criteria will fill out a personal information form and then be randomly assigned to groups using simple randomization method. Breathing exercises will be taught individually to participants in the experimental group by the researcher. In the experimental group, breathing exercises will be performed approximately 10 minutes, four times a day, starting from the first day after oral intake.
  Interventions: Behavioral: Breathing Exercise
- Control Group (No Intervention): No intervention other than routine nursing care will be performed.

INTERVENTIONS:
Behavioral: Breathing Exercise — He individual will be seated in a quiet environment in a semi-fowler or fowler position with their feet pointing forward. Then, they will be asked to join their hands on their abdomen and breathe normally while focusing on their breath. They will ensure their shoulders are relaxed, their body is loose, and they will inhale and exhale slowly and deeply through the nose without rushing.Next, while sitting upright with relaxed muscles, they will close their eyes, block their right nostril with their thumb or ring finger, inhale as much air as possible through the left nostril, and hold their breath. Then, they will block the left nostril with their ring finger or thumb and exhale slowly through the right nostril. The same process will be repeated for the left nostril. They will continue this process for approximately 2 minutes.
  Arms: Experimental Group

SUMMARY:
Surgical treatment is performed with the aim of reducing, halting the progression of, or treating certain pathological conditions in the human body by removing some tissue or organs from the body. Wedge resection is considered an effective method for the treatment of lung cancer. The wedge resection method is utilized in both malignant and non-malignant pulmonary pathologies (such as bronchiectasis, aspergilloma, non-tuberculous mycobacteria, tuberculosis, fungal infections, inflammatory pseudotumors, hydatid cyst, and benign masses). Following surgical procedures such as Video-Assisted Thorascopic Surgery (VATS) and wedge resection, side effects and complications such as atelectasis, pneumonia, acute respiratory distress syndrome, prolonged air leakage, chylothorax, sepsis, pneumothorax, pulmonary embolism, empyema, bronchopleural fistula, pain, anxiety, dyspnea, fatigue, and insomnia can occur.

Non-pharmacological methods are observed to increase comfort and control in patients, thereby enhancing their quality of life. Non-pharmacological interventions such as music therapy, hot or cold therapy, hypnosis, aromatherapy, massage, progressive relaxation exercises, deep breathing exercises, pursed lip breathing, yoga, and meditation can be employed in the management of postoperative symptoms such as pain, anxiety, dyspnea, insomnia, and fatigue. Studies involving breathing exercises have shown that they reduce anxiety and pain scores after exercise. Alternate nostril breathing, a yoga practice, is considered one of the best breathing exercises for health and fitness. It has positive effects on dyspnea, anxiety, stress, and sleep disorders.

DETAILED DESCRIPTION:
Surgical treatment is carried out with the aim of reducing, halting the progression of, or treating certain pathological conditions in the human body by removing some tissue or organs from the body. Wedge resection is considered an effective method for the treatment of lung cancer. The wedge resection method is utilized in both malignant and non-malignant pulmonary pathologies (such as bronchiectasis, aspergilloma, non-tuberculous mycobacteria, tuberculosis, fungal infections, inflammatory pseudotumors, hydatid cyst, and benign masses). Following surgical procedures such as VATS and wedge resection, side effects and complications such as atelectasis, pneumonia, acute respiratory distress syndrome, prolonged air leakage, chylothorax, sepsis, pneumothorax, pulmonary embolism, empyema, bronchopleural fistula, pain, anxiety, dyspnea, fatigue, and insomnia can occur.Non-pharmacological methods are observed to increase comfort and control in patients, thereby enhancing their quality of life. Non-pharmacological interventions such as music therapy, hot or cold therapy, hypnosis, aromatherapy, massage, progressive relaxation exercises, deep breathing exercises, pursed lip breathing, yoga, and meditation can be employed in the management of postoperative symptoms such as pain, anxiety, dyspnea, insomnia, and fatigue. Studies involving breathing exercises have shown that they reduce anxiety and pain scores after exercise. Alternate nostril breathing, a yoga practice, is considered one of the best breathing exercises for health and fitness. It has positive effects on dyspnea, anxiety, stress, and sleep disorders. Breathing exercises aim to improve individuals' quality of life and mitigate the effects of the disease, providing inexpensive and side-effect-free practices.Nurses should empower individuals to better manage symptoms such as experiencing less pain, reduced anxiety, alleviation or reduction of dyspnea, insomnia, fatigue, and other symptoms following surgical procedures. No study has been found that examines the effect of alternative nostril breathing exercises on pain, anxiety, dyspnea, fatigue, and insomnia symptoms in patients undergoing lung surgery. Our study aims to contribute to the literature by evaluating the effect of breathing exercises on pain, anxiety, dyspnea, and insomnia in patients undergoing lung resection and VATS procedures.Therefore, this study is planned to determine the effect of breathing exercises on pain, anxiety, dyspnea, and insomnia in patients undergoing lung resection and VATS procedures in a public hospital.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone VATS or wedge resection surgery,
* Having orientation to place and time,
* Being communicative,
* Having no visual or hearing impairment.

Exclusion Criteria:

* Having a mental health issue that would hinder communication,
* Having any nasal pathology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) - Pain Scale | First measurement on the day before surgery, second measurement on the first day after surgery, third measurement on the second day after surgery.
  A 10 cm ruler has been designed with painlessness on one side and the most severe pain possible on the other side. This ruler is known as the Visual Analog Scale (VAS) for visual comparison. In the evaluation of the scale, "0" indicates no pain, "1-3" indicates mild pain, "4-6" indicates moderate pain, and "7-10" indicates severe pain levels.
Visual Analog Scale (VAS) - Dyspnea Scale | First measurement on the day before surgery, second measurement on the first day after surgery, third measurement on the second day after surgery.
  The Visual Analog Scale (VAS) is applied by marking with a pencil on a horizontal or vertical line of one hundred millimeters. The 0 mm point of the line indicates no dyspnea, while the 100 mm point indicates the most severe dyspnea possible. The patient marks the severity of their current respiratory distress on the scale by using these two degrees as criteria.
State-Trait Anxiety Inventory | First measurement on the day before surgery, second measurement on the first day after surgery, third measurement on the second day after surgery.
  he development of the State-Trait Anxiety Inventory was conducted by Spielberger and his colleagues (1970), and it consists of two subscales: state anxiety and trait anxiety, each comprising 20 items. The scores obtained from both scales theoretically range between 20 and 80. A large score indicates a high level of anxiety, a small score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Richard Campbell Sleep Scale | First measurement on the day before surgery, second measurement on the first day after surgery, third measurement on the second day after surgery.
  It is a scale consisting of 6 items that assess the depth of nighttime sleep, the time it takes to fall asleep, the frequency of awakenings, the duration of wakefulness upon awakening, the quality of sleep, and the level of noise in the environment. Scores on the scale range from "0-25" indicating very poor sleep to "76-100" indicating very good sleep. While evaluating the total score of the scale based on 5 items, the 6th item, which assesses the level of noise in the environment, is excluded from the total score assessment. As the score on the scale increases, the quality of patients' sleep also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gündoğdu, PhD, Principal Investigator — KTO Karatay University; Hasibe Okutan, PhD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researcher at Konya City Hospital will collect the data.